CLINICAL TRIAL: NCT00998309
Title: Zithromax-SR 2g, Special Investigation For Skin And Soft Tissue Infection, Sexually-Transmitted Infection, And Infection Of The Oral (Regulatory Post Marketing Commitment Plan)
Brief Title: Zithromax-SR 2g, Special Investigation (Regulatory Post Marketing Commitment Plan)
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A0661202
Record Dates: First submitted 2009-10-16; First posted 2009-10-20 (Estimated); Results first posted 2012-05-01 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2012-04

CONDITIONS: Bacterial Infections
Keywords: skin infection; soft tissue infection; sexually-transmitted infection; infection oral; Regulatory Post Marketing Commitment Plan
MeSH Terms: conditions — Bacterial Infections; Cellulitis; Soft Tissue Infections; Sexually Transmitted Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Azithromycin SR: Patients taking Azithromycin.
  Interventions: Drug: Azithromycin SR

INTERVENTIONS:
Drug: Azithromycin SR — Zithromax SR 2g, taking once for treatment.
  Other Names: Zithromax SR, Azithromycin SR

SUMMARY:
To collect the efficacy and safety information of Zithromax-SR related to their appropriate use in daily practice.

DETAILED DESCRIPTION:
All the patients whom an investigator prescribes the first Azithromycin SR should be registered within 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects diagnosed with skin and soft tissue infection, sexually-transmitted infection, and infection of the oral.
* Subjects must have no prior experience with Azithromycin SR.

Exclusion Criteria:

* Patients not administered Azithromycin SR.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients whom an involving A0661202 prescribes the Azithromycin SR.
Sampling Method: Probability Sample
Enrollment: 502 (Actual)
Dates: Start 2009-10; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0661202&StudyName=Zithromax-SR%202g%2C%20Special%20Investigation%20%28Regulatory%20Post%20Marketing%20Commitment%20Plan%29%20

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a phase 4, observational, open-label study conducted in participants who were prescribed azithromycin by their treating physician per usual clinical practice. Study drug was not provided by the Sponsor.
Groups:
- Azithromycin SR: Azithromycin SR should be orally taken as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
Period: Overall Study
Arm/Group | Azithromycin SR
Started | 502
Completed | 498
Not Completed | 4
Not completed — Protocol Violation | 4

BASELINE CHARACTERISTICS:
Arm/Group | Azithromycin SR
Number analyzed (Participants) | 498
Age, Customized [Mean (Standard Deviation); unit: years] | 39.9 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 211
  Male | 287
Type of Infection [Number; unit: participants] — The physician in charge of the survey made the diagnosis of type of infection based on symptoms.
  participants
    Skin and Soft Tissue Infection | 104
    Sexual Transmitted Infection | 199
    Dental and Oral Surgery Infection | 183
    Others | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Investigator's Assessment of Clinical Outcome (Effective (Cured)/ Not Effective (Not Cured)) at End of the Study.
Description: The physician in charge of the survey performed comprehensive clinical effect evaluation on result of clinical findings, bacteriological effect and others. Clinical effect (Effective (cured)/ Not effective (not cured)/ unable to evaluate effectiveness evaluation) was performed at visits during the observation period by comparing to the data before administration of this drug.Criteria of cured was disappearance or improvement of clinical findings with infections and/or causal bacterial disappearance.
Time Frame: Baseline to 29 days
Population: The efficacy analysis population basically consists of the evaluable cases in accordance with the separately prepared analysis plan (cases judged to have been evaluated appropriately).
Measure: Number; unit: participants
Arm/Group | Azithromycin SR
Number analyzed (Participants) | 457
participants
  Effective (cured) | 438
  Not effective (not cured) | 19

2. Secondary Outcome: Risk Factors for the Proportion of Responders of Azithromycin (Clinical Effect)-Gender
Description: Number of participants with responders of azithromycin to determine whether male or female is significant risk factor.
Time Frame: Baseline to 29 days
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Azithromycin -Male: Male participants who took azithromycin SR orally as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
- Azithromycin-Female: Female Participants who took azithromycin SR orally as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
Arm/Group | Azithromycin -Male | Azithromycin-Female
Number analyzed (Participants) | 272 | 185
participants
  Number of participants | 272 | 185
  Participatns of Responders | 254 | 184
Statistical Analysis 1: Comparison: Azithromycin -Male vs Azithromycin-Female; The risk factor tested was "Gender". The null hypothesis is there is no difference between "males and females" in the participatns of responders; Test type: Superiority or Other; p = 0.001, Fisher Exact

3. Secondary Outcome: Risk Factors for the Proportion of Responders of Azithromycin (Clinical Effect)-Age
Description: Number of participants with responders of azithromycin to determine whether <65 years or >=65 years is significant risk factor.
Time Frame: Baseline to 29 days
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Azithromycin <65 Years: Participants with <65 years who took azithromycin SR as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
- Azithromycin->=65 Years: Participants>=65 years who took Azithromycin SR as a single dose of 2 g (potency, as azithromycin) with an empty stomach according to Japanese Package Insert.
Arm/Group | Azithromycin <65 Years | Azithromycin->=65 Years
Number analyzed (Participants) | 414 | 43
participants
  Number of participants | 414 | 43
  Participatns of Responders | 396 | 42
Statistical Analysis 1: Comparison: Azithromycin <65 Years vs Azithromycin->=65 Years; The risk factor tested was "Age". The null hypothesis is there is no difference between "<65 years and >=65 years " in the participatns of responders; Test type: Superiority or Other; p = 1.000, Fisher Exact

4. Secondary Outcome: Risk Factors for the Proportion of Responders of Azithromycin (Clinical Effect)-Type of Infection
Description: Number of participants with responders of azithromycin to determine whether type of infection, "Skin and Soft Tissue Infection, Sexual Transmitted Infection, or Dental and Oral Surgery Infection", is significant risk factor.
Time Frame: Baseline to 29 days
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Azithromycin -Skin and Soft Tissue Infection: Participants with Skin and Soft Tissue Infection (SSTI) who took azithromycin SR as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
- Azithromycin-Sexual Transmitted Infection: Participants with Sexual Transmitted Infection (STI) who took azithromycin SR as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
- Aazithromycin-Dental and Oral Surgery Infection: Participants with Dental and Oral Surgery Infection (DOSI) who took azithromycin SR as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
Arm/Group | Azithromycin -Skin and Soft Tissue Infection | Azithromycin-Sexual Transmitted Infection | Aazithromycin-Dental and Oral Surgery Infection
Number analyzed (Participants) | 96 | 199 | 162
participants
  Number of participants | 96 | 199 | 162
  Participatns of Responders | 95 | 181 | 162
Statistical Analysis 1: Comparison: Azithromycin -Skin and Soft Tissue Infection vs Azithromycin-Sexual Transmitted Infection vs Aazithromycin-Dental and Oral Surgery Infection; The risk factor tested was "type of infection". The null hypothesis is there is no difference amang "Skin and Soft Tissue Infection, Sexual Transmitted Infection, and Dental and Oral Surgery Infection" in the participatns of responders; Test type: Superiority or Other; p < 0.001, Fisher Exact

5. Secondary Outcome: Risk Factors for the Proportion of Responders of Azithromycin (Clinical Effect)-Infection Severity
Description: Number of participants with responders of azithromycin to determine whether Infection severity, "mild infection, moderate infection, or severe infection", is significant risk factor.
Time Frame: Baseline to 29 days
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Azithromycin-mild Infection: Participants with mild infection who took azithromycin SR as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
- Azithromycin-moderate Infection: Participants with moderate infection who took azithromycin SR as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
  , moderate infection, or severe in
- Azithromycin-severe Infection: Participants with severe infection who took azithromycin SR as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
Arm/Group | Azithromycin-mild Infection | Azithromycin-moderate Infection | Azithromycin-severe Infection
Number analyzed (Participants) | 152 | 260 | 45
participants
  Number of Participants | 152 | 260 | 45
  Participatns of Responders | 147 | 247 | 44
Statistical Analysis 1: Comparison: Azithromycin-mild Infection vs Azithromycin-moderate Infection vs Azithromycin-severe Infection; The risk factor tested was "Infection severity". The null hypothesis is there is no difference amang "mild infection, moderate infection, and severe infection" in the participatns of responders; Test type: Superiority or Other; p = 0.556, Fisher Exact

6. Secondary Outcome: Risk Factors for the Proportion of Responders of Azithromycin (Clinical Effect)-Hepatic Dysfunction(HD)
Description: Number of participants with responders of azithromycin to determine whether with or without hepatic dysfunction is significant risk factor.
Time Frame: Baseline to 29 days
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Azithromycin -Without Hepatic Dysfunction: Participants without Hepatic Dysfunction (HD) who took azithromycin SR as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
- Azithromycin-with Hepatic Dysfunction: Participants with Hepatic Dysfunction (HD) who took azithromycin SR as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
Arm/Group | Azithromycin -Without Hepatic Dysfunction | Azithromycin-with Hepatic Dysfunction
Number analyzed (Participants) | 395 | 2
participants
  Number of Participants | 395 | 2
  Participatns of Responders | 381 | 1
Statistical Analysis 1: Comparison: Azithromycin -Without Hepatic Dysfunction vs Azithromycin-with Hepatic Dysfunction; The risk factor tested was "hepatic dysfunction". The null hypothesis is there is no difference between "with and without hepatic dysfunction" in the participatns of responders; Test type: Superiority or Other; p = 0.074, Fisher Exact

7. Secondary Outcome: Risk Factors for the Proportion of Responders of Azithromycin (Clinical Effect)-Renal Dysfunction(RD)
Description: Number of participants with responders of azithromycin to determine whether with or without renal dysfunction is significant risk factor.
Time Frame: Baseline to 29 days
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Azithromycin-without Renal Dysfunction: Participants without Renal Dysfunction (RD) who took azithromycin SR as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
- Azithromycin-with Renal Dysfunction: Participants with Renal Dysfunction (RD) who took azithromycin SR as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
Arm/Group | Azithromycin-without Renal Dysfunction | Azithromycin-with Renal Dysfunction
Number analyzed (Participants) | 397 | 1
participants
  Number of Participants | 397 | 1
  Participatns of Responders | 382 | 1
Statistical Analysis 1: Comparison: Azithromycin-without Renal Dysfunction vs Azithromycin-with Renal Dysfunction; The risk factor tested was "Renal dysfunction". The null hypothesis is there is no difference between "with and without Renal dysfunction" in the participatns of responders; Test type: Superiority or Other; p = 1.000, Fisher Exact

8. Secondary Outcome: Risk Factors for the Proportion of Responders of Azithromycin (Clinical Effect)-Past Medical History (PMH)
Description: Number of participants with responders of azithromycin to determine whether with or without past medical history is significant risk factor.
Time Frame: Baseline to 29 days
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Azithromycin-without Past Medical History: Participants without Past Medical History (PMH) who took azithromycin SR as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
- Azithromycin- With Past Medical History: Participants with Past Medical History (PMH) who took azithromycin SR as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
Arm/Group | Azithromycin-without Past Medical History | Azithromycin- With Past Medical History
Number analyzed (Participants) | 441 | 16
participants
  Number of Participants | 441 | 16
  Participatns of Responders | 422 | 16
Statistical Analysis 1: Comparison: Azithromycin-without Past Medical History vs Azithromycin- With Past Medical History; The risk factor tested was "Past medical history". The null hypothesis is there is no difference between "with and without past medical history" in the participatns of responders; Test type: Superiority or Other; p = 1.000, Fisher Exact

9. Secondary Outcome: Risk Factors for the Proportion of Responders of Azithromycin (Clinical Effect)-Complications
Description: Number of participants with responders of azithromycin to determine whether with or without complications is significant risk factor.
Time Frame: Baseline to 29 days
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Azithromycin Without Complications: Participants without Complications who took azithromycin SR as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
- Azithromycin With Complications: Participants with Complications who took azithromycin SR as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
Arm/Group | Azithromycin Without Complications | Azithromycin With Complications
Number analyzed (Participants) | 408 | 49
participants
  Number of Participants | 408 | 49
  Participatns of Responders | 391 | 47
Statistical Analysis 1: Comparison: Azithromycin Without Complications vs Azithromycin With Complications; The risk factor tested was "complications". The null hypothesis is there is no difference between "with and without complications " in the participatns of responders; Test type: Superiority or Other; p = 1.000, Fisher Exact

10. Secondary Outcome: Risk Factors for the Proportion of Responders of Azithromycin (Clinical Effect)-Previous Antibiotic Treatment History (PATH)
Description: Number of participants with responders of azithromycin to determine whether with or without previous antibiotic treatment history is significant risk factor.
Time Frame: Baseline to 29 days
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Azithromycin Without PATH: Participants without Previous Antibiotic Treatment History (PATH) who took azithromycin SR as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
- Azithromycin With PATH: Participants with Previous Antibiotic Treatment History (PATH) who took azithromycin SR as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
Arm/Group | Azithromycin Without PATH | Azithromycin With PATH
Number analyzed (Participants) | 441 | 16
participants
  Number of Participants | 441 | 16
  Participatns of Responders | 422 | 16
Statistical Analysis 1: Comparison: Azithromycin Without PATH vs Azithromycin With PATH; The risk factor tested was "previous antibiotic treatment history". The null hypothesis is there is no difference between "with and without previous antibiotic treatment history" in the participatns of responders; Test type: Superiority or Other; p = 1.000, Fisher Exact

11. Secondary Outcome: Risk Factors for the Proportion of Responders of Azithromycin (Clinical Effect)-Comcomittant Drugs(CD)
Description: Number of participants with responders of azithromycin to determine whether with or without comcomittant drugs is significant risk factor.
Time Frame: Baseline to 29 days
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Azithromycin Without Comcomittant Drugs: Participants without Comcomittant Drugs (CD) who took azithromycin SR as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
- Azithromycin With Comcomittant Drugs: Participants with Comcomittant Drugs (CD) who took azithromycin SR as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
Arm/Group | Azithromycin Without Comcomittant Drugs | Azithromycin With Comcomittant Drugs
Number analyzed (Participants) | 284 | 173
participants
  Number of Participants | 284 | 173
  Participatns of Responders | 274 | 164
Statistical Analysis 1: Comparison: Azithromycin Without Comcomittant Drugs vs Azithromycin With Comcomittant Drugs; The risk factor tested was "comcomittant drugs". The null hypothesis is there is no difference between "with and without comcomittant drugs" in the participatns of responders; Test type: Superiority or Other; p = 0.470, Fisher Exact

12. Secondary Outcome: Risk Factors for the Proportion of Responders of Azithromycin (Clinical Effect)-Non-Drug Therapy
Description: Number of participants with responders of azithromycin to determine whether with or without non-drug therapy is significant risk factor.
Time Frame: Baseline to 29 days
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Azithromycin -With Non-Drug Therapy: Participants without Non-Drug Therapy who took azithromycin SR as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
- Azithromycin-with Non-Drug Therapy: Participants with Non-Drug Therapy who took azithromycin SR as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
Arm/Group | Azithromycin -With Non-Drug Therapy | Azithromycin-with Non-Drug Therapy
Number analyzed (Participants) | 423 | 34
participants
  Number of Participants | 423 | 34
  Participatns of Responders | 405 | 33
Statistical Analysis 1: Comparison: Azithromycin -With Non-Drug Therapy vs Azithromycin-with Non-Drug Therapy; The risk factor tested was "non-drug therapy". The null hypothesis is there is no difference between "with and without non-drug therapy" in the participatns of responders; Test type: Superiority or Other; p = 1.000, Fisher Exact

13. Primary Outcome: Number of Participants With Treatment Related Adverse Events (TRAEs)
Description: All observed or volunteered adverse events and the investigator's opinion of the causal relationship to the study treatment were reported. Defenition of an adverse event (AE) is any adverse change in health or side effect that occurs in participates. Treatment related Adverse Events were evaluated in company with the causal relationship to the investigational product.
Time Frame: Baseline to 29 days
Population: The safety analysis population consists of the cases that satisfy the paticipants conditions and in whom administration of this drug was confirmed.
Measure: Number; unit: participants
Arm/Group | Azithromycin SR
Number analyzed (Participants) | 498
participants
  Number of Participants without TRAEs | 446
  Number of Participants with TRAEs | 52

14. Primary Outcome: Number of Unlisted Treatment Related Adverse Events (TRAEs)
Description: All observed or volunteered adverse events and the investigator's opinion of the causal relationship to the study treatment were reported. Defenition of an adverse event (AE) is any adverse change in health or side effect that occurs in participates. Treatment related Adverse Events were evaluated in company with the causal relationship to the investigational product. Unlisted treatment related adverse events were confirmed with listed adverse drug reaction in Japanese package insert.
Time Frame: Baseline to 29 days
Population: as for outcome 13
Measure: Number; unit: Events
Arm/Group | Azithromycin SR
Number analyzed (Participants) | 498
Events
  Number of Treatment Related AEs Analyzed | 61
  Number of Unlisted Treatment Related AEs | 2

15. Secondary Outcome: Risk Factors for Incidence Rate of Treatment Related Adverse Events (TRAEs) of Azithromycin -Gender
Description: Number of participants with Treatment Related Adverse Events (TRAEs) of azithromycin to determine whether male or female is significant risk factor.
Time Frame: Baseline to 29 days
Population: as for outcome 13
Measure: Number; unit: participants
Groups:
- Azithromycin Male: Male participants who took azithromycin SR as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
- Azithromycin Female: Female participants who took azithromycin SR as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
Arm/Group | Azithromycin Male | Azithromycin Female
Number analyzed (Participants) | 287 | 211
participants
  Number of Participants | 287 | 211
  Number of Participants with TRAEs | 32 | 20
Statistical Analysis 1: Comparison: Azithromycin Male vs Azithromycin Female; The risk factor tested was "Gender". The null hypothesis is there is no difference between "males and females" in the Incidence Rate of Treatment Related Adverse Events (TRAEs); Test type: Superiority or Other; p = 0.657, Fisher Exact

16. Secondary Outcome: Risk Factors for Incidence Rate of Treatment Related Adverse Events (TRAEs) of Azithromycin -Age
Description: Number of participants with Treatment Related Adverse Events (TRAEs) of azithromycin to determine whether <65 years or >=65 years is significant risk factor.
Time Frame: Baseline to 29 days
Population: as for outcome 13
Measure: Number; unit: participants
Groups:
- Azithromycin <65 Years: Participants <65 years who took azithromycin SR as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
- Azithromycin >=65 Years: Participants >=65 years who took azithromycin SR as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
Arm/Group | Azithromycin <65 Years | Azithromycin >=65 Years
Number analyzed (Participants) | 448 | 50
participants
  Number of Participants | 448 | 50
  Number of Participants with TRAEs | 50 | 2
Statistical Analysis 1: Comparison: Azithromycin <65 Years vs Azithromycin >=65 Years; The risk factor tested was "Age". The null hypothesis is there is no difference between "<65 years or >=65" in the Incidence Rate of Treatment Related Adverse Events (TRAEs); Test type: Superiority or Other; p = 0.145, Fisher Exact

17. Secondary Outcome: Risk Factors for Incidence Rate of Treatment Related Adverse Events (TRAEs) of Azithromycin -Type of Infection
Description: Number of participants with Treatment Related Adverse Events (TRAEs) of azithromycin to determine whether Type of Infection, "Skin and Soft Tissue Infection, Sexual Transmitted Infection, or Dental, or Oral Surgery Infection", is significant risk factor.
Time Frame: Baseline to 29 days
Population: as for outcome 13
Measure: Number; unit: participants
Groups:
- Azithromycin - Skin and Soft Tissue Infection: Participants with Skin and Soft Tissue Infection who took azithromycin SR as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
- Azithromycin - Sexual Transmitted Infection: Participants with "Skin and Soft Tissue Infection, Sexual Transmitted Infection, or Dental, or Oral Surgery Infection"who took azithromycin SR as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
- Azithromycin-Dental, or Oral Surgery Infection: Participants with Dental, or Oral Surgery Infection who took azithromycin SR as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
Arm/Group | Azithromycin - Skin and Soft Tissue Infection | Azithromycin - Sexual Transmitted Infection | Azithromycin-Dental, or Oral Surgery Infection
Number analyzed (Participants) | 104 | 199 | 183
participants
  Number of Participants | 104 | 199 | 183
  Number of Participants with TRAEs | 2 | 24 | 26
Statistical Analysis 1: Comparison: Azithromycin - Skin and Soft Tissue Infection vs Azithromycin - Sexual Transmitted Infection vs Azithromycin-Dental, or Oral Surgery Infection; The risk factor tested was "Type of Infection". The null hypothesis is there is no difference amang "Skin and Soft Tissue Infection, Sexual Transmitted Infection, and Dental or Oral Surgery Infection" in the Incidence Rate of Treatment Related Adverse Events (TRAEs); Test type: Superiority or Other; p = 0.005, Fisher Exact

18. Secondary Outcome: Risk Factors for Incidence Rate of Treatment Related Adverse Events (TRAEs) of Azithromycin -Infection Severity
Description: Number of participants with Treatment Related Adverse Events (TRAEs) of azithromycin to determine whether mild infection, moderate infection, or severe infection is significant risk factor.
Time Frame: Baseline to 29 days
Population: as for outcome 13
Measure: Number; unit: participants
Groups:
- Azithromycin-moderate Infection: Participants with moderate infection who took azithromycin SR as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
Arm/Group | Azithromycin-mild Infection | Azithromycin-moderate Infection | Azithromycin-severe Infection
Number analyzed (Participants) | 168 | 283 | 47
participants
  Number of Participants | 168 | 283 | 47
  Number of Participants with TRAEs | 19 | 25 | 8
Statistical Analysis 1: Comparison: Azithromycin-mild Infection vs Azithromycin-moderate Infection vs Azithromycin-severe Infection; The risk factor tested was "Infection severity". The null hypothesis is there is no difference amang "mild infection, moderate infection, or severe infection" in the Incidence Rate of Treatment Related Adverse Events (TRAEs); Test type: Superiority or Other; p = 0.213, Fisher Exact

19. Secondary Outcome: Risk Factors for Incidence Rate of Treatment Related Adverse Events (TRAEs) of Azithromycin -Hepatic Dysfunction
Description: Number of participants with Treatment Related Adverse Events (TRAEs) of azithromycin to determine whether with or without Hepatic Dysfunction is significant risk factor.
Time Frame: Baseline to 29 days
Population: as for outcome 13
Measure: Number; unit: participants
Groups:
- Azithromycin Without Hepatic Dysfunction: Participants without Hepatic Dysfunction who took azithromycin SR as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
- Azithromycin With Hepatic Dysfunction: Participants with Hepatic Dysfunction who took azithromycin SR as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
Arm/Group | Azithromycin Without Hepatic Dysfunction | Azithromycin With Hepatic Dysfunction
Number analyzed (Participants) | 422 | 2
participants
  Number of Participants | 422 | 2
  Number of Participants with TRAEs | 48 | 0
Statistical Analysis 1: Comparison: Azithromycin Without Hepatic Dysfunction vs Azithromycin With Hepatic Dysfunction; The risk factor tested was "Hepatic Dysfunction". The null hypothesis is there is no difference between "with and without Hepatic Dysfunction" in the Incidence Rate of Treatment Related Adverse Events (TRAEs); Test type: Superiority or Other; p = 1.000, Fisher Exact

20. Secondary Outcome: Risk Factors for Incidence Rate of Treatment Related Adverse Events (TRAEs) of Azithromycin -Renal Dysfunction
Description: Number of participants with Treatment Related Adverse Events (TRAEs) of azithromycin to determine whether with or without Renal Dysfunction is significant risk factor.
Time Frame: Baseline to 29 days
Population: as for outcome 13
Measure: Number; unit: participants
Groups:
- Azithromycin Without Renal Dysfunction: Participants without Renal Dysfunction who took azithromycin SR as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
- Azithromycin- With Renal Dysfunction: Participants with Renal Dysfunction who took azithromycin SR as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
Arm/Group | Azithromycin Without Renal Dysfunction | Azithromycin- With Renal Dysfunction
Number analyzed (Participants) | 423 | 1
participants
  Number of Participants | 423 | 1
  Number of Participants with TRAEs | 48 | 1
Statistical Analysis 1: Comparison: Azithromycin Without Renal Dysfunction vs Azithromycin- With Renal Dysfunction; The risk factor tested was "Renal Dysfunction". The null hypothesis is there is no difference between "with and without Renal Dysfunction" in the Incidence Rate of Treatment Related Adverse Events (TRAEs); Test type: Superiority or Other; p = 0.116, Fisher Exact

21. Secondary Outcome: Risk Factors for Incidence Rate of Treatment Related Adverse Events (TRAEs) of Azithromycin -Past Medical History
Description: Number of participants with Treatment Related Adverse Events (TRAEs) of azithromycin to determine whether with or without Past Medical History is significant risk factor.
Time Frame: Baseline to 29 days
Population: as for outcome 13
Measure: Number; unit: participants
Groups:
- Azithromycin -Without Past Medical History: Participants without Past Medical History who took azithromycin SR as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
- Azithromycin- With Past Medical History: Participants with Past Medical History who took azithromycin SR as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
Arm/Group | Azithromycin -Without Past Medical History | Azithromycin- With Past Medical History
Number analyzed (Participants) | 481 | 17
participants
  Number of Participants | 481 | 17
  Number of Participants with TRAEs | 42 | 10
Statistical Analysis 1: Comparison: Azithromycin -Without Past Medical History vs Azithromycin- With Past Medical History; The risk factor tested was "Past Medical History". The null hypothesis is there is no difference between "with and without Past Medical History" in the Incidence Rate of Treatment Related Adverse Events (TRAEs); Test type: Superiority or Other; p < 0.001, Fisher Exact

22. Secondary Outcome: Risk Factors for Incidence Rate of Treatment Related Adverse Events (TRAEs) of Azithromycin -Complications
Description: Number of participants with Treatment Related Adverse Events (TRAEs) of azithromycin to determine whether with or without complications is significant risk factor.
Time Frame: Baseline to 29 days
Population: as for outcome 13
Measure: Number; unit: participants
Groups:
- Azithromycin -Without Complications: Participants without complications who took azithromycin SR as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
- Azithromycin-with Complications: Participants with complications who took azithromycin SR as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
Arm/Group | Azithromycin -Without Complications | Azithromycin-with Complications
Number analyzed (Participants) | 441 | 57
participants
  Number of Participants | 441 | 57
  Number of Participants with TRAEs | 45 | 7
Statistical Analysis 1: Comparison: Azithromycin -Without Complications vs Azithromycin-with Complications; The risk factor tested was "complications". The null hypothesis is there is no difference between "with and without complications" in the Incidence Rate of Treatment Related Adverse Events (TRAEs); Test type: Superiority or Other; p = 0.645, Fisher Exact

23. Secondary Outcome: Risk Factors for Incidence Rate of Treatment Related Adverse Events (TRAEs) of Azithromycin -Previous Antibiotic Treatment History (PATH)
Description: Number of participants with Treatment Related Adverse Events (TRAEs) of azithromycin to determine whether with or without previous antibioutic treatment history (PATH) is significant risk factor.
Time Frame: Baseline to 29 days
Population: as for outcome 13
Measure: Number; unit: participants
Groups:
- Azithromycin Without PATH: Participants without previous antibioutic treatment history (PATH) who took azithromycin SR as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
- Azithromycin-with PATH: Participants with previous antibioutic treatment history (PATH) who took azithromycin SR as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
Arm/Group | Azithromycin Without PATH | Azithromycin-with PATH
Number analyzed (Participants) | 481 | 16
participants
  Number of Participants | 481 | 16
  Number of Participants with TRAEs | 50 | 2
Statistical Analysis 1: Comparison: Azithromycin Without PATH vs Azithromycin-with PATH; The risk factor tested was "previous antibiotic treatment history (PATH)". The null hypothesis is there is no difference between "with and without previous antibiotic treatment history (PTH)" in the Incidence Rate of Treatment Related Adverse Events (TRAEs); Test type: Superiority or Other; p = 0.679, Fisher Exact

24. Secondary Outcome: Risk Factors for Incidence Rate of Treatment Related Adverse Events (TRAEs) of Azithromycin -Comcomittant Drugs
Description: Number of participants with Treatment Related Adverse Events (TRAEs) of azithromycin to determine whether with or without comcomittant drugs is significant risk factor.
Time Frame: Baseline to 29 days
Population: as for outcome 13
Measure: Number; unit: participants
Groups:
- Azithromycin Without Comcomittant Drugs: Participants without comcomittant drugs who took azithromycin SR as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
- Azithromycin- With Comcomittant Drugs: Participants with comcomittant drugs who took azithromycin SR as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
Arm/Group | Azithromycin Without Comcomittant Drugs | Azithromycin- With Comcomittant Drugs
Number analyzed (Participants) | 298 | 200
participants
  Number of Participants | 298 | 200
  Number of Participants with TRAEs | 27 | 25
Statistical Analysis 1: Comparison: Azithromycin Without Comcomittant Drugs vs Azithromycin- With Comcomittant Drugs; The risk factor tested was "comcomittant drugs". The null hypothesis is there is no difference between "with and without comcomittant drugs" in the Incidence Rate of Treatment Related Adverse Events (TRAEs); Test type: Superiority or Other; p = 0.234, Fisher Exact

25. Secondary Outcome: Risk Factors for Incidence Rate of Treatment Related Adverse Events (TRAEs) of Azithromycin -Non-Drug Therapy
Description: Number of participants with Treatment Related Adverse Events (TRAEs) of azithromycin to determine whether with or without non-drug therapy is significant risk factor.
Time Frame: Baseline to 29 days
Population: as for outcome 13
Measure: Number; unit: participants
Groups:
- Azithromycin Without Non-drug Therapy: Participants without non-drug therapy who took azithromycin SR as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
- Azithromycin With Non-drug Therapy: Participants with non-drug therapy who took azithromycin SR as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
Arm/Group | Azithromycin Without Non-drug Therapy | Azithromycin With Non-drug Therapy
Number analyzed (Participants) | 463 | 35
participants
  Number of Participants | 463 | 35
  Number of Participants with TRAEs | 52 | 0
Statistical Analysis 1: Comparison: Azithromycin Without Non-drug Therapy vs Azithromycin With Non-drug Therapy; The risk factor tested was "non-drug therapy". The null hypothesis is there is no difference between "with and without non-drug therapy" in the Incidence Rate of Treatment Related Adverse Events (TRAEs); Test type: Superiority or Other; p = 0.039, Fisher Exact

26. Secondary Outcome: Risk Factors for Incidence Rate of Treatment Related Adverse Events (TRAEs) of Azithromycin -Pregnancy in Female
Description: Number of participants with Treatment Related Adverse Events (TRAEs) of azithromycin to determine whether with or without Pregnancy in Female is significant risk factor.
Time Frame: Baseline to 29 days
Population: as for outcome 13
Measure: Number; unit: participants
Groups:
- Azithromycin Without Pregnancy in Female: Female participants without Pregnancy who took azithromycin SR as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
- Azithromycin With Pregnancy in Female: Female participants with Pregnancy who took azithromycin SR as a single dose of 2 g with an empty stomach according to Japanese Package Insert.
Arm/Group | Azithromycin Without Pregnancy in Female | Azithromycin With Pregnancy in Female
Number analyzed (Participants) | 199 | 11
participants
  Number of Participants | 199 | 11
  Number of Participants with TRAEs | 20 | 0
Statistical Analysis 1: Comparison: Azithromycin Without Pregnancy in Female vs Azithromycin With Pregnancy in Female; The risk factor tested was "Pregnancy" in Female. The null hypothesis is there is no difference between "with and without Pregnancy" in the Incidence Rate of Treatment Related Adverse Events (TRAEs) in Female; Test type: Superiority or Other; p = 0.605, Fisher Exact

ADVERSE EVENTS:
Description: The frequency of treatment related adverse events during the study.
Arm/Group | Azithromycin SR
Serious Adverse Events (participants affected / at risk) | 0/498
Other Adverse Events (participants affected / at risk) | 52/498
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azithromycin SR (N=498)
Diarrhea (Gastrointestinal disorders) | 44 (44)
Nausea (Gastrointestinal disorders) | 4 (4)
Enterocolitis (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (3)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Face Oedema (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.